CLINICAL TRIAL: NCT02805127
Title: Obstructive Airways Diseases in Emergency Department (OADED) Study
Status: Terminated | Type: Observational
Why Stopped: Lower recruitment rate than expected
Sponsor: Oridion (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Organization: Medtronic - MITG (Industry)
Other Study IDs: MDT17071
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Asthma; COPD; Capnography
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with COPD and Asthma .: Patients with COPD and Asthma. Continuous capnography and spirometry measurements of the subjects will be taken form the subjects with at least two minutes recording before the first spirometry assessment.
  All clinical diagnoses and treatments will be performed according to the department's protocols.
  This is an observational study with no interventions

SUMMARY:
This is an observational study which aims to evaluate the possibility of using data from a capnography device to assess obstructive airway severity in both Chronic Obstructive Pulmonary Disease (COPD) and Asthma patients.

DETAILED DESCRIPTION:
This is a feasibility observational study which aims to evaluate the possibility of using data from a capnography device to assess obstructive airway severity in both COPD and Asthma patients. The study will include adults asthma and COPD patients (age >18) that arrive at the Emergency Department (ED). Patients will be enrolled on a continuous basis and will be monitored by a capnograph and an oximeter before, during and after lung function assessment and medical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Ability and willingness to participate the study and sign informed consent form
3. Asthma / COPD patients

Exclusion Criteria:

1. Pregnant women
2. Asthma or COPD patients with FEV1 > 60%
3. Disability or unwillingness to undergo capnography measurement
4. Cannot be assessed for FEV1
5. Oxygen supply >5 L/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma and COPD patients
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-12-22; Primary Completion 2017-08-06 (Actual); Study Completion 2017-08-06 (Actual)

PRIMARY OUTCOMES:
Correlation between capnography parameters and severity of asthma | 1/2 hour to 48 hours from enrollment of subjects
  Correlation between the airway obstruction severity calculation based on the capnography parameters and the clinical severity of asthma and COPD as defined by forced expiratory volume in 1 second (FEV1), in severe asthma and COPD patients

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Stalnikowicz, Prof. ; M.D., Principal Investigator — Emergency Department, Hadassah University Hospital Mount Scopus

IPD SHARING:
Plan to Share IPD: No